CLINICAL TRIAL: NCT07008170
Title: Laparoendoscopic Rendezvous for Difficult Cholecystocholedocholithiasis.
Brief Title: Laparoendoscopic Rendezvous for Concomitant Gall Bladder Stones and Common Bile Duct Stones
Acronym: LERV
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Minia University (Other)
Responsible Party: Principal Investigator, Saleh Khairy Saleh MD, Lecturer, Minia University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1379/12/2024
Record Dates: First submitted 2025-05-28; First posted 2025-06-06 (Actual); Last update posted 2025-06-19 (Actual); Status verified 2025-06

CONDITIONS: Gall Stone; Common Bile Duct Calculi; Cholecystitis, Chronic; Choledocholithiasis; Periampullary Diverticula
MeSH Terms: conditions — Gallstones; Cholecystitis; Bronchiolitis Obliterans Syndrome; Choledocholithiasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Laparoendoscopic rendezvous(LERV) (Other): Step 1: Laparoscopic Phase Step 2: Endoscopic Phase Step 3: Completion
  Interventions: Procedure: Laparoendoscopic rendezvous

INTERVENTIONS:
Procedure: Laparoendoscopic rendezvous — The main principles of LERV technique consists of
  1. An antegrade trans cystic cannulation of the bile duct during laparoscopic cholecystectomy, with a guidewire that can be retrieved with a duodenoscope, thus facilitating retrograde bile duct cannulation.
  2. An over-the-wire sphincterotome is then inserted and standard maneuvers of endoscopic common bile duct stones clearance are performed.
  3. The procedure is then completed by cholecystectomy in one procedure

SUMMARY:
Chronic calculous cholecystitis in pediatric patients leads to choledocholithiasis in about 12% of cases. These patients require removal of stones from the common bile duct. The most common method of cleaning the common bile duct is endoscopic retrograde cholangiopancreatography, and the standard technique for removing the gallbladder is laparoscopic cholecystectomy. There are different approaches to the treatment of this category of patients: laparoscopic common bile duct exploration (LCBDE), laparoendoscopic rendezvous method (LERV) and one-stage LC( laparoscopic cholecystectomy) after ERCP( endoscopic retrograde cholangiopancreatography).

The aim of this prospective study is to evaluate the efficacy and safety Laparoendoscopic rendezvous for difficult cholecystocholedocholithiasis.

DETAILED DESCRIPTION:
The incidence of concomitant choledocholithiasis in patients with gallstone disease has been reported to range between 10% and 20% depending on geographic distribution.The ideal management of cholecysto-choledocholithiasis is still a matter of debate; different modalities, including the open and the laparoscopic approach, and sequential or simultaneous techniques, have been applied with success.

The management of gallbladder stones (lithiasis) concomitant with bile duct stones is controversial. The management of CBD( common bile duct) stones has evolved considerably since the advent of laparoscopic surgery. The more frequent approach is a two-stage procedure, with endoscopic sphincterotomy and stone removal from the bile duct followed by laparoscopic cholecystectomy. The laparoscopic-endoscopic rendezvous combines the two techniques in a single-stage operation. So the aim of this study was to evaluate one-stage LC with intra-operative endoscopic sphincterotomy (IOES) vs two-stage pre-operative endoscopic sphincterotomy (POES) followed by LC for the treatment of cholecystocholedocholithiasis Endoscopic Retrograde Cholangiopancreatography (ERCP) is one of the most technically challenging procedures in gastrointestinal endoscopy. Selective deep cannulation is a critical step for the performance of ERCP. The incidence of difficult cannulation has been reported in many studies, ranging from 10% to 40% in patients with native papilla. Difficult cannulation is an independent risk factor for post-ERCP pancreatitis (PEP).

The definition of difficult cannulation has been proposed by European Society of Gastrointestinal Endoscopy (ESGE) guidelines. Initial cannulation is considered difficult with the presence of one or more of the following: more than 5 min for attempting to cannulate; more than 5 contacts with the papilla; more than 1 unintended pancreatic duct cannulation or opacification.

Aim of the study is to evaluate use of laparoendoscopic rendezvous for difficult cholecystocholedocholithiasis using preprocedural abdominal CT findings. Primary outcome is to performs difficult biliary cannulation by rendezvous technique while secondary outcomes is to to detect morbidity (especially post-ERCP pancreatitis) , success of CBD clearance and to detect overall hospital

Risk factors of difficult cannulation during ERCP based on preprocedural abdominal CT findings in the study :

1. periampullary diverticulum
2. Location of the major papilla other than the descending duodenum
3. Presence of papilla bulging
4. Choledochoduodenal (CD) angle: the angle between the distal common bile duct and adjacent duodenum,
5. CBD( common bile duct) diameter
6. Far distal CBD (common bile duct) stone B. Laboratory investigation: normal bilirubin C. Previous upper gastrointestinal tract surgery/ Surgically altered anatomy

ELIGIBILITY:
Inclusion Criteria:

* Patients having stone(s) in the gallbladder and concurrent common bile duct , as determined by MRCP(magnetic resonance cholangiopancreatography) or US.
* Patients with acute cholecystitis, acute cholangitis, obstructive jaundice, and those with highly suspicious criteria for common bile duct stones, such as dilated CBD( common bile duct ) on US examination > 7 mm in diameter without obvious common bile duct stones, high serum bilirubin level, and/or high serum alkaline phosphatase level, were also included in this study. (high risk for cholecystocholedocholithiasis)
* Previous failed ERCP attempt
* Patients fit for general anesthesia and tolerant of pneumoperitoneum and endoscopic procedures.

Exclusion Criteria:

* History of hepatobiliary surgery as choledochoduodenal anastomosis
* A Previous upper abdominal surgery as total or partial gastric resection.
* Morbid obesity.
* Uncorrectable coagulopathy.
* Patients who refused to give consent.
* Pregnancy.
* Suspected malignant biliary stricture or cholangiocarcinoma
* Severe acute cholangitis with hemodynamic instability or septic shock requiring immediate biliary drainage (may necessitate emergent ERCP or percutaneous drainage first)
* Impacted CBD stones or stones deemed too large for endoscopic extraction (e.g., > 1.5 cm)
* Severe cardiopulmonary disease significantly increasing operative risk.
* Intrahepatic bile duct stones with indications for surgery.
* Patients with choledocholithiasis >2 cm or a large number of stones were difficult to remove.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-06-15 (Actual); Primary Completion 2026-06-15 (Estimated); Study Completion 2026-07-15 (Estimated)

PRIMARY OUTCOMES:
Assess the success rate of LERV for difficult cannulation | Intraoperative
  Assess the success rate of LERV for difficult cannulation

SECONDARY OUTCOMES:
assess the success rate of LERV in clearing the common bile duct in patients with choledocholithiasis | intraoperative
  CBD clearance success,Complete extraction of all stones during LERV judged by ERCP imaging
incidence of postsphincterotomy bleeding | 30 days after LERV
  obvious bleeding during ERCP Or delayed as melena
incidence of Acute pancreatitis | 30 days after ERCP
  increase serum amylase and lipase
Recurrence of common bile duct stones | 60 days after LERV
  The diagnosis of the stone in the common bile duct was made by MRI, CT scan and ultrasound.
Incidence of bile leak | 30 days after LERV
  bile aspirated from the abdominal cavity
incidence of Perforation | 30 days after LERV
  by CT, radiography (fluid or gas in the retroperitoneal space or abdominal cavity, visual picture during endoscopic examination)
incidence of Acute cholangitis | 60 days after LERV
  intermittent chills, fever, increased proinflammatory blood markers after ERCP
incidence of bile duct stricture | 1 year after LERV
  after LERV

CONTACTS AND LOCATIONS:
Overall Officials: Saleh K Saleh, MD, Principal Investigator — Minia University
Locations (1):
- Liver and GIT hospital , Minia University, Minya, Egypt

IPD SHARING:
Plan to Share IPD: No